CLINICAL TRIAL: NCT03709381
Title: Effect of Adrenocorticotropic Hormone on Vascular Endothelial Growth Factor Release in Healthy Children and Adolescent
Brief Title: Effect of Adrenocorticotropic Hormone on Vascular Endothelial Growth Factor Release in Children Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryan Heksch, Fellow, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB17-00194
Record Dates: First submitted 2017-10-02; First posted 2018-10-17 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Adrenal Insufficiency; Osteopenia, Osteoporosis; Steroid Suppression of ACTH Secretion
Keywords: steroid-induced adrenal suppression; vascular endothelial growth factor; adrenocorticotropic hormone; osteopenia
MeSH Terms: conditions — Adrenal Insufficiency; Bone Diseases, Metabolic | interventions — Cosyntropin; Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: At t=0, 9 ml of blood will be collected for measurement of VEGF, ACTH, and cortisol levels. Then, 1 mcg of cosyntropin (a synthetic ACTH analog) will be administered intravenously (IV). Samples for measurement of cortisol and VEGF levels will be obtained at t=30 and 60 minutes (6 ml of blood collected at both times). After the 60 minute blood draw, 250 mcg of cosyntropin will be administered IV. At t=90, 120, 150 , and 180 minutes, samples for measurement of cortisol and VEGF levels will be obtained (6 ml of blood collected at each time).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACTH stim test arm (Experimental): Cosyntropin 1 mcg IV (low dose) will be given to subjects at t=0 minutes, and Cosyntropin 250 mcg (high dose) IV will be given to subjects at t=60 minutes. (All subjects were in the same arm and had the same protocol).
  Interventions: Drug: Low Dose Cosyntropin (ACTH) stimulation test; Drug: High Dose Cosyntropin (ACTH) stimulation test

INTERVENTIONS:
Drug: Low Dose Cosyntropin (ACTH) stimulation test — Cosyntropin 1 mcg IV given to subjects at t=0
Drug: High Dose Cosyntropin (ACTH) stimulation test — Cosyntropin 250 mcg IV given to subjects at t=60

SUMMARY:
Bone disease and adrenal suppression are two of the many side effects of steroid use in pediatrics. Evidence has shown that adrenocorticotropic hormone (ACTH) protects against the adverse bone effects of steroids in animals and in vitro models, but this has not yet been evaluated in humans. The proposed mechanism in these studies is that ACTH stimulates osteoblasts in bone to release Vascular Endothelial Growth Factor (VEGF), which increases the vascularity in high risk areas of bone. This can potentially be protective against osteonecrosis and osteopenia, which can lead to bone fractures if not prevented. The VEGF release can also be used to demonstrate that an administration of exogenous ACTH occurred. This could be important in diagnosing adrenal insufficiency (AI). One of the tests to assess central AI is the low-dose ACTH stimulation test (LDAST). This test has a high rate of false positive results due to technical limitations. However, if an ACTH-stimulated VEGF level can be measured during the test as a marker of the test being done properly, it will allow for proper interpretation of the results (and identification of a false positive), which will reduce the number of patients being incorrectly diagnosed with central AI.

This study will recruit ten healthy children and adolescents, ages 9-18, to assess the effects of ACTH on VEGF levels. The investigators will measure the response of VEGF and cortisol to an administration of a low dose and high dose of cosyntropin (the synthetic ACTH analog used in this test). The hypothesis of this study is that VEGF and cortisol will both increase after administration of cosyntropin. At this time, no other studies have demonstrated that VEGF is responsive to ACTH in humans. If the hypothesis is correct, the results will have two main implications. VEGF can be used as a marker of ACTH administration during the LDAST to identify false positive tests. Secondly, this will help further research into whether ACTH can be used to protect against bone disease in high-dose steroid-treated patients. Further studies can be done to assess whether this effect will be the same in patients with AI or steroid-induced adrenal suppression.

DETAILED DESCRIPTION:
Problem: Chronic steroid use causes a wide range of side effects, of which bone disease and adrenal suppression cause significant morbidity. Bone disease, which includes osteopenia, fractures, and osteonecrosis, is very common. In patients on chronic steroids, fractures can occur in up to 30-50%, low bone mineral density (BMD) can occur in up to 50%, and up to 40% have some degree of osteonecrosis. Another common side effect of steroid use is suppression of the HPA axis. This can cause a patient's endogenous cortisol and ACTH production to be reduced, which can take up to several months to return to baseline after discontinuing steroids. Diagnosing adrenal suppression can be difficult. Literature exists showing that ACTH can stimulate release of VEGF (in vitro and in animal in vivo studies), which can both be protective against bone disease and be used as a marker of exogenous cosyntropin administration. The primary goal of this study is to show that ACTH can increase VEGF levels in healthy humans.

Bone disease: As stated above, patients taking chronic steroids are at high risk for significant bone effects. Glucocorticoids cause osteoblast apoptosis and decreased function while simultaneously decreasing apoptosis of osteoclasts, overall resulting in decreased bone formation and higher resorption. This leads to low BMD and fractures. Osteonecrosis can also be due to glucocorticoid causing decreased angiogenesis in high risk areas of bone (i.e. the femoral head). In rabbits,one study demonstrated that ACTH use protects against osteonecrosis by stimulating osteoblasts to release VEGF, which maintains good blood flow to these high risk areas of bone. Another study demonstrated that Cushing Syndrome patients with ACTH-producing pituitary tumors had less BMD loss than those with adrenal cortisol-producing tumors. This outcome points toward ACTH being protective against osteopenia (even in a high steroid state). The mechanism for this protective effect is unclear but could be through ACTH stimulation of VEGF. It is unknown whether ACTH increases VEGF in humans and if it does the dose needed and timeframe of the response need to be determined.

Low-dose ACTH stimulation test (LDAST): There are several methods to evaluate adrenal insufficiency (AI), however the LDAST is best for diagnosing central AI and steroid-induced adrenal suppression (SIAS). The Metyrapone test is very specific, but it carries the risk of causing acute AI and requires a hospitalization to administer. The insulin tolerance test is the gold standard for diagnosing AI, but also carries the risk of causing hypoglycemia. The "standard" or high-dose (250mcg) ACTH stimulation test is a good test as well for diagnosing primary AI, but can result in false negatives that miss patients with central AI or SIAS, which can have significant morbidity (sensitivity for central AI is only 73%). Primary AI can also be diagnosed with an elevated ACTH level, but central AI and SIAS usually have a low to normal ACTH. Therefore, the LDAST test was created to help increase the rate of patients with central AI being diagnosed, with a sensitivity for central AI at 93%. However, there are several limitations to the LDAST. Cosyntropin is dispensed in 250 mcg vials, which is used for the high-dose test. and must be diluted to 1 mcg for the LDAST. The medication also runs the risk of sticking to IV tubing. Therefore, it is occasionally not truly given to the patient, which can cause a false positive result (the lack of cortisol response to ACTH is not due to AI, but due to never receiving cosyntropin). Due to these limitations, the specificity for diagnosing central AI is 90%. This can cause the interpreting physician to diagnose AI, and prescribe a hydrocortisone, when the patient did not truly have AI.

If the LDAST had a positive control to show that the cosyntropin appropriately reached the patient, it would help to allow the endocrinologist to recognize a false positive result. As stated above, VEGF is stimulated by ACTH in animals. If VEGF levels were measured with cortisol levels, and they rose above a set threshold, the interpreting physician could feel more comfortable knowing that the test was administered appropriately. For VEGF to be a good control value, it would need to have a significant rise in response to cosyntropin, and would need to rise quickly and after one dose (the LDAST lasts one hour) and be independent of the cortisol response. In the in vitro study above, steroid-treated cells had significant rise in VEGF within one hour of ACTH treatment, and VEGF stayed elevated for up to four hours. In a study looking at whether VEGF could be a diagnostic biomarker to differentiate acute stroke in adults versus stroke mimics, there was a significant elevation of VEGF at the time of stroke presentation compared to the average normal value (peak median 1700 pg/mL with interquartile range of 1500-1900; baseline median 466 with interquartile range of 392-649). The mechanism for rise in VEGF was postulated to be due to a hypoxia stimulus in this case. However, it seems that VEGF can be acutely stimulated (potentially within one hour of a stimulus) and has the ability to rise to several standard deviations above the normal median baseline value in humans.

VEGF: Vascular Endothelial Growth Factor is a cytokine glycoprotein that is responsible for angiogenesis, or the formation of new blood vessels. It can also maintain blood vessel density, thickness, and permeability, and it is vital for endothelial cell survival. VEGF is a family of cytokines, with VEGF-A being the prototype and most common. It is found in the lungs, kidneys, heart, adrenals, bone, brain, and several other organs. Within the adrenal, VEGF has been shown to be stimulated by ACTH and can be protective against atrophy in steroid use. Important in regards to this study, an animal study showed that VEGF can be stimulated by ACTH outside the adrenal glands, namely in osteoblasts in bone. Osteoblasts have an MC2R receptor that is stimulated by ACTH, leading to a rise in VEGF levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 9-18 years old on the day of testing

Exclusion Criteria:

* Currently taking any medication other than over-the-counter medications (over-the-counter medications will be stopped on the day of the study)
* Steroid use within the prior six months (including IV, oral, inhaled, and intranasal steroids)
* Oral Contraceptive Pill use within the prior six months
* Any chronic medical conditions
* Pregnancy

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Difference between VEGF levels at baseline and the peak VEGF level after low dose cosyntropin administration in healthy children and adolescents | From t=0 minutes to t=60 minutes (1 hour total)
  Prior to administering Cosyntropin, a VEGF level will be obtained. 1 mcg Cosyntropin will be administered at t=0, then VEGF will be measured at 30 and 60 minutes. The investigators will run a comparison on the peak plasma VEGF level (the higher of the 30 and 60 minute level) after low dose stimulation compared to baseline VEGF levels.

SECONDARY OUTCOMES:
Difference between VEGF levels at baseline and the peak VEGF level after high dose cosyntropin administration in healthy children and adolescents | From t=60 minutes to t=180 minutes (2 hours total)
  After the 60 minute blood draw, a high dose (250 mcg) of Cosyntropin will be given. VEGF levels will be obtained every 30 minutes for another 2 hours (t=90, 120,150,180 min). The investigators will run a comparison on the peak plasma VEGF level (the highest of the 90, 120,150,180 minute levels) after high dose stimulation compared to baseline VEGF levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Heksch, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD